CLINICAL TRIAL: NCT04225767
Title: Phase II Investigation of Calcium Electroporation as a Treatment for Cutaneous and Subcutaneous Malignant Tumours
Brief Title: Calcium Electroporation as a Treatment for Cutaneous and Subcutaneous Malignant Tumours
Acronym: CaEP-R
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: Vejle Hospital (Other); University College Absalon (Other); University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REG-115-2019
Record Dates: First submitted 2019-12-27; First posted 2020-01-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Cancer
Keywords: Calcium; Electroporation; Cancer; Skin
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Calcium electroporation treatment (Experimental): Experimental treatment with calcium electroporation for malignant cutaneous and subcutaneous tumours
  Interventions: Combination Product: Calcium electroporation

INTERVENTIONS:
Combination Product: Calcium electroporation — Patients with cutaneous or subcutaneous malignant tumours will be treated with calcium electroporation, i.e. intratumoral injection of calcium followed by electroporation by electric pulses applied directly to the tumor.

SUMMARY:
Phase II Investigation of Calcium Electroporation as a Treatment for Cutaneous and Subcutaneous Malignant Tumours.

DETAILED DESCRIPTION:
This will be a non-randomized phase II trial with the objective of evaluating the clinical response rate of calcium electroporation treatment of malignant tumours of the skin and assessing treatment impact on quality of life. This study will investigate the response rate of calcium electroporation treatment of skin metastases and malignant wounds in a real-world setting, in three different cancer centres in Northern Europe. The centres aim to treat a total of 30 patients with cancer in the skin of any histology. The patients will be treated once and followed with regular examinations for 12 months, starting from first treatment day. All patients will have been offered the standard of care and all available alternatives before entering the protocol. Calcium electroporation will not be compared to other means of treatment.

The primary endpoint of this study is to evaluate the clinical overall response rate of calcium electroporation treatment of malignant tumours of the skin after two months. A subset of patients will undergo MR scans after treatment and another subset of patients will be interviewed regarding treatment impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Trial subject ≥ 18 years.
* Trial subject must be able to understand the participant information.
* Histologically verified cutaneous or subcutaneous, primary or secondary cancer of any histology.
* The patient must have been offered other relevant standard treatment for their cancer disease.
* The patient can undergo any simultaneous medical treatment (endocrine therapy, chemotherapy, immunotherapy etc.) if progressive or stable disease is present after a treatment period of two months or more.
* The patient can undergo radiation therapy, provided that the treatment field does not involve treated area.
* Performance status ECOG/WHO ≤2.
* At least one cutaneous or subcutaneous tumour measuring up to 3 cm.
* Both men and women who are sexually active must use safe contraception (contraceptive coil, deposit injection of gestagen, subdermal implantation, hormonal vaginal ring or transdermal patch).
* Signed informed consent.

Exclusion Criteria:

• Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Tumour response (size) | 2 months
  Response rate will be defined as number of responding lesions (partial or complete response) relative to treated lesions evaluated by changes in size (mm) by clinical examination with caliper measurement. Tumor response will be further documented using clinical photography.

SECONDARY OUTCOMES:
Treatment response up to 12 months (size) | 13 months
  Evaluate treatment response at month 1, 3, 4, 6 and 12 in addition to evaluating treatment response after 2 months. Response rate will be defined as number of responding lesions (partial or complete response) relative to treated lesions evaluated by changes in size (mm) by clinical examination with caliper measurement. Tumor response will be further documented using clinical photography.
Assessment of residual tumor from biopsies after 1 year | 12 months
  Assess tumour and surrounding tissue response to treatment from biopsies of the treated area after 1 year. Microscopy assessment of histopathological regressive changes (eg. % tumor cells and fibrosis).
MRI scans to verify treatment and evaluate tumour changes after treatment | 2 months
  Assess response after treatment on MRI scans on a subset of patients before and immediately after treatment, as well as after 2 months using diffusion-weighted magnetic resonance imaging (DW-MRI) as a method to monitor electroporated tissue, using the concept of the apparent diffusion coefficient (ADC).
Evaluation of patient quality of life before and after treatment using EORTC Questionnaires. | 13 months
  Evaluate patient quality of life before treatment, after 2 months and after 1 year through EORTC QLQ-C15-PAL Core questionnaires evaluating cancer-related symptoms on a scale from 1-4 (not at all-very much) as well as overall quality of life on a scale from 1-7 (very poor-excellent).
Systemic immunologic response evaluated by routine scans | 12 months
  Investigate any sign of systemic immunologic response from any routine scans (MRI, PET-CT etc.) before and after treatment in the inclusion period by tumor size and TNM stage.
Response according to tumour histology | 12 months
  To list response rates and response duration according to tumour histology.
Remission | 12 months
  To determine complete and partial remissions for all tumours treated. Response rate will be defined as number of responding lesions (partial or complete response) relative to treated lesions evaluated by changes in size (mm) by clinical examination with caliper measurement. Tumor response will be further documented using clinical photography.
Individual response | 12 months
  To determine rate of response for each individual patient.
Importance of irradiation | 12 months
  To investigate response (overall, as well as complete and partial) depending whether the treated tumour was in a previously irradiated area. Response rate will be defined as number of responding lesions (partial or complete response) relative to treated lesions evaluated by changes in size (mm) by clinical examination with caliper measurement. Tumor response will be further documented using clinical photography.
Current measurement | 1 day
  To measure current during treatment as measured by the pulse generator.
Evaluation of changes in quality of life through qualitative interview | 2 months
  Analyses of qualitative interviews (in a subset of patients) performed before- and 2 months after treatment that include measures related to patient experience and impact on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gehl, MD, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vissing M, Ploen J, Pervan M, Vestergaard K, Schnefeldt M, Frandsen SK, Rafaelsen SR, Lindhardt CL, Jensen LH, Rody A, Gehl J. Study protocol designed to investigate tumour response to calcium electroporation in cancers affecting the skin: a non-randomised phase II clinical trial. BMJ Open. 2021 Jun 16;11(6):e046779. doi: 10.1136/bmjopen-2020-046779. PMID 34135049